CLINICAL TRIAL: NCT02797171
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Pharmacokinetics, and Anti-Viral Activity of VRC-HIVMAB060-00-AB (VRC01) and VRC-HIVMAB080-00-AB (VRC01LS) in the Serum and Mucosa of Healthy, HIV-Uninfected Adult Participants
Brief Title: Evaluating the Safety, Pharmacokinetics, and Anti-Viral Activity of VRC01 and VRC01LS in the Serum and Mucosa of Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 116; 20733 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): Participants will receive 10 mg/kg of VRC01 at Months 0, 2, 4, and 6.
  Interventions: Biological: VRC01
- Group 2 (Experimental): Participants will receive 30 mg/kg of VRC01 at Months 0, 2, 4, and 6.
  Interventions: Biological: VRC01
- Group 3 (Experimental): Participants will receive 30 mg/kg of VRC01LS at Months 0, 3, and 6.
  Interventions: Biological: VRC01LS
- Group 4 (Experimental): Participants will receive 30 mg/kg of VRC01 at Month 0.
  Interventions: Biological: VRC01
- Group 5 (Experimental): Participants will receive 30 mg/kg of VRC01LS at Month 0.
  Interventions: Biological: VRC01LS

INTERVENTIONS:
Biological: VRC01 — Administered by intravenous (IV) infusion
  Other Names: VRC-HIVMAB060-00-AB
  Arms: Group 1; Group 2; Group 4
Biological: VRC01LS — Administered by intravenous (IV) infusion
  Other Names: VRC-HIVMAB080-00-AB
  Arms: Group 3; Group 5

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and antiviral activity of VRC-HIVMAB060-00-AB (VRC01) and VRC-HIVMAB080-00-AB (VRC01LS) in the serum and mucosa of healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate two experimental human monoclonal antibodies (mAbs): VRC-HIVMAB060-00-AB (VRC01) and VRC-HIVMAB080-00-AB (VRC01LS). VRC01LS is designed to have a longer half-life than VRC01. The purpose of this study is to evaluate the safety, pharmacokinetics, and antiviral activity of VRC01 and VRC01LS in the serum and mucosa of healthy, HIV-uninfected adults.

This study will enroll healthy, HIV-uninfected adults into five groups. At various time points during the study, participants in Groups 1, 2, and 4 will receive intravenous (IV) infusions of VRC01, and participants in Groups 3 and 5 will receive IV infusions of VRC01LS. Participants in Groups 1, 2, and 3 will attend 13 to 14 study visits over about 1 to 1 ½ years; participants in Groups 4 and 5 will attend 7 to 9 study visits over about 6 months to 1 year. At certain time points, study visits will include physical examinations, blood collection, urine collection, and interviews and questionnaires. At other time points, depending on group assignment and gender, visits will also include collection of cervicovaginal secretions, rectal secretions, and semen; and cervical, vaginal, and rectal biopsies.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria:

* Age of 18 to 50 years
* Weight less than or equal to 115 kg
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to enrollment with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until completion of the last study visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection [low risk guidelines are found on the protocol home page on the HVTN Members' site (https://members.hvtn.org/protocols/hvtn116)] and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit

Laboratory Inclusion Values:

Hemogram/CBC

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 2,500 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: U.S. volunteers must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA). Non-U.S. sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range)

Reproductive Status:

* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to initial biopsy for groups 1-3 and prior to initial infusion for groups 4-5 on the day of enrollment. Persons who are NOT of reproductive potential due to having undergone bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.

Reproductive Status:

United States:

A volunteer who was born female must:

* Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:

  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception, or
  * Any other contraceptive method approved by the HVTN 116 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
* Or not be of reproductive potential, such as having had a bilateral oophorectomy, or tubal ligation;
* Or be sexually abstinent.

South Africa:

A volunteer who was born female must:

* Agree to consistently use effective contraception (see the protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in South Africa is defined as using 2 methods of birth control.

ONE barrier contraceptive method:

* Condoms (male or female)
* Diaphragm or cervical cap

PLUS ONE of the following methods:

* Intrauterine device (IUD),
* Hormonal contraception, or
* Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy), or
* Any other contraceptive method approved by the HVTN 116 PSRT

Or not be of reproductive potential, such as having had a bilateral oophorectomy, or tubal ligation;

Or be sexually abstinent.

* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Mucosal Specimen Collection

* Volunteers 21 years of age and older who were born female: Pap smear (verified by medical records) is required within:

  * the 3 years prior to enrollment with the latest result reported as normal or ASCUS (atypical squamous cells of undetermined significance), OR
  * the 5 years prior to enrollment, with the latest result reported as normal, or ASCUS with no evidence of high risk HPV.
  * If no Pap smear was done within the last 3 years (or within the last 5 years, if high risk HPV testing was performed), the volunteer must be willing to undergo a Pap smear with the result reported (verified by medical records) as normal or ASCUS prior to sample collection.
* Willing to have mucosal secretions and tissue biopsies collected
* Willing to abstain from sexual intercourse for the required period after each biopsy collection

Exclusion Criteria:

General

* Blood products received within 120 days before first infusion, unless eligibility for earlier enrollment is determined by the HVTN 116 PSRT
* Investigational research agents received within 30 days before first infusion
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 116 study
* Pregnant or breastfeeding
* Active duty U.S. military personnel with the potential of being deployed during the study

Vaccines and Other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 116 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 6 months in a prior vaccine trial. Exceptions may be made for some vaccines and vaccine trials. For volunteers who have received an experimental vaccine(s) less than 6 months ago, eligibility for enrollment will be determined by the HVTN 116 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 10 days before first infusion or scheduled within 10 days after first infusion (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Previous receipt of humanized or human mAbs whether licensed or investigational

Immune System

* Immunosuppressive medications received within 30 days before first infusion. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; or [3] topical corticosteroids for mild, uncomplicated dermatitis)
* Serious adverse reactions to VRC01 and VRC01LS formulation components such as sodium citrate, sodium chloride, and L-arginine hydrochloride, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain
* Autoimmune disease (Not exclusionary: mild, well-controlled psoriasis)
* Immunodeficiency

Clinically Significant Medical Conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated infusions or blood draws, including perceived inability to establish venous access
  * A condition that requires regular use of any anticoagulant medications (not including aspirin or NSAIDs),
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to study product, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

  * Exclude a volunteer who:
  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease unless well controlled (normal T3/T4/TSH) with medication
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* For those undergoing rectal biopsies, a rectal condition, such as an active infection or inflammation of the colorectal area (e.g., an HSV-2 outbreak or inflamed hemorrhoids or colitis/diarrhea), internal hemorrhoids, or any other condition noted during screening rectal exam via anoscope or in medical history that in the opinion of the clinician represents a contraindication to mucosal sampling
* For those undergoing vaginal and cervical biopsies, any condition noted during pelvic exam via speculum or in medical history that in the opinion of the clinician represents a contraindication to mucosal sampling
* An active genital tract condition, such as an active infection or inflammation of the genital tract (e.g., genital sores or ulcers, penile or abnormal vaginal discharge, genital warts that are symptomatic or requiring treatment) or any other condition that in the opinion of the clinician represents a contraindication to mucosal sampling
* Hysterectomy
* Menopause

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie McElrath, Study Chair — Seattle Vaccine Trials Unit; Linda-Gail Bekker, Study Chair — Desmond Tutu HIV Centre
Locations (4):
- United States (3):
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Groote Schuur HIV CRS, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Lemos MP, Astronomo RD, Huang Y, Narpala S, Prabhakaran M, Mann P, Paez CA, Lu Y, Mize GJ, Glantz H, Westerberg K, Colegrove H, Smythe KS, Lin M, Pierce RH, Hutter J, Frank I, Mascola JR, McDermott AB, Bekker LG, McElrath MJ. Enhanced and sustained biodistribution of HIV-1 neutralizing antibody VRC01LS in human genital and rectal mucosa. Nat Commun. 2024 Nov 28;15(1):10332. doi: 10.1038/s41467-024-54580-9. PMID 39609400

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: VRC01 10 mg/kg mo(0,2,4,6)
- Group 2: Vaccine: VRC01 30 mg/kg mo(0,2,4,6)
- Group 3: Vaccine: VRC01LS 30 mg/kg mo(0,3,6)
- Group 4: Vaccine: VRC01 30 mg/kg mo(0)
- Group 5: Vaccine: VRC01LS 30 mg/kg mo(0)
- Group 6: Pre-treatment: Biopsy collected but was not randomized to any treatment group
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Started | 23 | 23 | 7 | 16 | 10 | 1
Safety Population | 23 | 23 | 7 | 16 | 10 | 1
Completed | 19 | 21 | 5 | 15 | 8 | 0
Not Completed | 4 | 2 | 2 | 1 | 2 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant unable to adhere | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Not Randomized | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: In Groups 1-3, participants who have their biopsies collected at visit 2; in Groups 4-5, participants who receive infusion at visit 3
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment | Total
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1 | 80
Age, Continuous [Median (Full Range); unit: years] | 31 [22 to 47] | 27 [21 to 50] | 33 [23 to 43] | 30 [18 to 39] | 30 [21 to 41] | 34 [34 to 34] | 29 [18 to 50]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 0 | 0 | 0 | 2 | 0 | 0 | 2
  21 - 30 years | 11 | 16 | 3 | 7 | 5 | 0 | 42
  31 - 40 years | 7 | 5 | 3 | 7 | 4 | 1 | 27
  41 - 50 years | 5 | 2 | 1 | 0 | 1 | 0 | 9
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 3 | 8 | 6 | 0 | 43
  Male | 10 | 10 | 4 | 8 | 4 | 1 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 22 | 23 | 7 | 16 | 10 | 1 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 12 | 5 | 4 | 1 | 1 | 35
  White | 9 | 6 | 2 | 11 | 8 | 0 | 36
  More than one race | 1 | 3 | 0 | 1 | 1 | 0 | 6
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 13 | 12 | 3 | 16 | 10 | 0 | 54
  South Africa | 10 | 11 | 4 | 0 | 0 | 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017] The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after each infusion at months 0, 2, 3, 4 or 6 (infusion visits depending on which group participants are in)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10
Participants
  Pain: None | 19 | 18 | 7 | 15 | 10
  Pain: Mild | 4 | 5 | 0 | 1 | 0
  Pain: Moderate | 0 | 0 | 0 | 0 | 0
  Pain: Severe | 0 | 0 | 0 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Tenderness: None | 19 | 16 | 7 | 13 | 9
  Tenderness: Mild | 4 | 6 | 0 | 3 | 1
  Tenderness: Moderate | 0 | 1 | 0 | 0 | 0
  Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 18 | 15 | 7 | 13 | 9
  Pain and/or Tenderness: Mild | 5 | 7 | 0 | 3 | 1
  Pain and/or Tenderness: Moderate | 0 | 1 | 0 | 0 | 0
  Pain and/or Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: None | 22 | 21 | 7 | 16 | 10
  Erythema/Redness: Mild | 0 | 2 | 0 | 0 | 0
  Erythema/Redness: Moderate | 1 | 0 | 0 | 0 | 0
  Erythema/Redness: Severe | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 22 | 23 | 7 | 16 | 10
  Induration/Swelling: Mild | 1 | 0 | 0 | 0 | 0
  Induration/Swelling: Moderate | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Severe | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 22 | 21 | 7 | 16 | 10
  Erythema and/or Induration: Mild | 0 | 2 | 0 | 0 | 0
  Erythema and/or Induration: Moderate | 1 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10
Participants
  Malaise and/or fatigue: None | 14 | 18 | 6 | 12 | 9
  Malaise and/or fatigue: Mild | 7 | 3 | 1 | 3 | 1
  Malaise and/or fatigue: Moderate | 2 | 2 | 0 | 1 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 21 | 19 | 7 | 15 | 9
  Myalgia: Mild | 2 | 4 | 0 | 1 | 1
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Headache: None | 13 | 17 | 7 | 15 | 10
  Headache: Mild | 9 | 4 | 0 | 0 | 0
  Headache: Moderate | 1 | 2 | 0 | 1 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Nausea: None | 20 | 19 | 5 | 14 | 10
  Nausea: Mild | 3 | 4 | 1 | 2 | 0
  Nausea: Moderate | 0 | 0 | 1 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Vomiting: None | 22 | 22 | 5 | 16 | 10
  Vomiting: Mild | 1 | 1 | 2 | 0 | 0
  Vomiting: Moderate | 0 | 0 | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Chills: None | 21 | 23 | 7 | 16 | 10
  Chills: Mild | 1 | 0 | 0 | 0 | 0
  Chills: Moderate | 1 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 22 | 22 | 7 | 15 | 10
  Arthralgia: Mild | 1 | 1 | 0 | 1 | 0
  Arthralgia: Moderate | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Diarrhea: None | 20 | 17 | 7 | 15 | 10
  Diarrhea: Mild | 2 | 6 | 0 | 1 | 0
  Diarrhea: Moderate | 1 | 0 | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0 | 0 | 0
  Diarrhea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 10 | 14 | 3 | 11 | 8
  Max. Systemic Symptoms: Mild | 11 | 7 | 3 | 4 | 2
  Max. Systemic Symptoms: Moderate | 2 | 2 | 1 | 1 | 0
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Temperature: None | 21 | 22 | 7 | 16 | 10
  Temperature: Mild | 2 | 1 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Chemistry and Hematology Laboratory Measures
Description: alkaline phosphate (ALP) (U/L), aspartate aminotransferase (AST) (U/L), alanine aminotransferase (ALT) (U/L) (Doesn't mention about lab grade > 1 )
Time Frame: Measured through IV infusion at visits 1 (screening), 4 (day 1-15), 7 (day 57-71), 10 (day 99-113), 12 (day 127-141), 14 (day 169-183), 16 (day 252-267), and 18 (day 442-456) (visits depending on which group participants are in)
Population: Visit schedule is not the same for each treatment group. For visits not on the schedule, number analyzed is 0 and median/IQR is ---.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1
U/L
  ALT (SGPT) (U/L)- Screening | 16 [13 to 22] | 16 [12 to 22] | 17 [12 to 25] | 15.5 [12 to 21] | 13 [9 to 15] | 33 [33 to 33]
  ALT (SGPT) (U/L)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  ALT (SGPT) (U/L)- Day 1 - 15 | 15 [12 to 23] | 15 [11 to 20] | 21 [15 to 22] | 13 [10.5 to 19.5] | 13.5 [10 to 26] |
  ALT (SGPT) (U/L)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 57 - 71 | 15 [11 to 20] | 16 [15 to 19] |  |  |  |
  ALT (SGPT) (U/L)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 99 - 113 |  |  | 22 [14 to 37] |  |  |
  ALT (SGPT) (U/L)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  ALT (SGPT) (U/L)- Day 127 - 141 | 15.5 [11.5 to 20.5] | 18.5 [13.5 to 23] |  | 13 [9 to 16] |  |
  ALT (SGPT) (U/L)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 169 - 183 | 16 [12.5 to 20] | 15.5 [11 to 18.5] | 17 [13 to 26] |  |  |
  ALT (SGPT) (U/L)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 1 | 0 | 8 | 0
  ALT (SGPT) (U/L)- Day 252 - 267 | 15.5 [13 to 22.5] | 19 [13 to 23] | 25 [25 to 25] |  | 18.5 [13.5 to 37] |
  ALT (SGPT) (U/L)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 442 - 456 |  |  | 19 [11 to 57] |  |  |
  AST (U/L)- Screening | 20 [17 to 22] | 20 [18 to 23] | 22 [17 to 27] | 19 [16.5 to 21] | 15.5 [13 to 19] | 32 [32 to 32]
  AST (U/L)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  AST (U/L)- Day 1 - 15 | 19 [17 to 22] | 20 [18 to 23] | 22 [18 to 37] | 18 [16 to 21] | 19.5 [15 to 30] |
  AST (U/L)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  AST (U/L)- Day 57 - 71 | 18 [17 to 22] | 19 [17 to 24] |  |  |  |
  AST (U/L)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  AST (U/L)- Day 99 - 113 |  |  | 25 [16 to 40] |  |  |
  AST (U/L)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  AST (U/L)- Day 127 - 141 | 19.5 [16.5 to 23] | 21 [17 to 25] |  | 17 [14 to 20] |  |
  AST (U/L)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  AST (U/L)- Day 169 - 183 | 19 [17 to 22] | 20.5 [17 to 24] | 20 [19 to 40] |  |  |
  AST (U/L)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  AST (U/L)- Day 252 - 267 | 18.5 [16.5 to 21.5] | 20 [17 to 24] |  |  | 19 [13.5 to 27.5] |
  AST (U/L)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  AST (U/L)- Day 442 - 456 |  |  | 17 [16 to 39] |  |  |
  Alkaline Phosphatase (U/L)- Screening | 65 [58 to 85] | 61 [49 to 69] | 71 [60 to 87] | 52.5 [46 to 60.5] | 55.5 [55 to 73] | 97 [97 to 97]
  Alkaline Phosphatase (U/L)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Alkaline Phosphatase (U/L)- Day 1 - 15 | 65 [61 to 73] | 60 [53 to 70] | 69 [63 to 80] | 54 [45.5 to 62] | 60.5 [58 to 74] |
  Alkaline Phosphatase (U/L)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 57 - 71 | 67 [61 to 74] | 67 [55 to 77] |  |  |  |
  Alkaline Phosphatase (U/L)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 99 - 113 |  |  | 72 [62 to 86] |  |  |
  Alkaline Phosphatase (U/L)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 127 - 141 | 68 [61 to 77.5] | 67.5 [55 to 80] |  | 52 [45 to 65] |  |
  Alkaline Phosphatase (U/L)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 169 - 183 | 68.5 [61 to 83.5] | 63 [54.5 to 72.5] | 79.5 [71 to 89] |  |  |
  Alkaline Phosphatase (U/L)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Alkaline Phosphatase (U/L)- Day 252 - 267 | 68 [56.5 to 83] | 59 [52 to 68] |  |  | 70.5 [56 to 96.5] |
  Alkaline Phosphatase (U/L)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 442 - 456 |  |  | 70 [69 to 101] |  |  |

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine, Hemoglobin
Description: Chemistry and Hematology Laboratory Measures - creatinine (g/dl), hemoglobin (g/dl)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1
g/dl
  Hemoglobin (g/dL)- Screening | 14.5 [13.4 to 15] | 14 [13 to 15.2] | 13.7 [13.7 to 16.6] | 14.75 [12.95 to 15.35] | 13.3 [12.4 to 14.9] | 14.9 [14.9 to 14.9]
  Hemoglobin (g/dL)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Hemoglobin (g/dL)- Day 1 - 15 | 13.8 [13.1 to 14.6] | 13.3 [12.3 to 14.5] | 13.7 [12.6 to 15.2] | 14 [12.65 to 15.1] | 12.95 [11.9 to 15] |
  Hemoglobin (g/dL)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 57 - 71 | 14.1 [12.8 to 14.4] | 14 [12.6 to 14.5] |  |  |  |
  Hemoglobin (g/dL)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 99 - 113 |  |  | 14.6 [12.5 to 15.6] |  |  |
  Hemoglobin (g/dL)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Hemoglobin (g/dL)- Day 127 - 141 | 13.7 [12.7 to 14.5] | 13.25 [12.45 to 14.75] |  | 14.3 [12.9 to 15.9] |  |
  Hemoglobin (g/dL)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 169 - 183 | 14 [12.9 to 14.35] | 13 [12.2 to 14.8] | 13.7 [12.7 to 16] |  |  |
  Hemoglobin (g/dL)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Hemoglobin (g/dL)- Day 252 - 267 | 14.05 [13.2 to 14.4] | 13.4 [12.3 to 14.9] |  |  | 14.25 [12.8 to 14.6] |
  Hemoglobin (g/dL)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 442 - 456 |  |  | 14.6 [13.4 to 15.7] |  |  |
  Creatinine (g/dL)- Screening | 0.00073 [0.00062 to 0.00082] | 0.00074 [0.0006 to 0.00083] | 0.00071 [0.0007 to 0.00085] | 0.00085 [0.00074 to 0.00091] | 0.00074 [0.0007 to 0.00089] | 0.00086 [0.00086 to 0.00086]
  Creatinine (g/dL)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Creatinine (g/dL)- Day 1 - 15 | 0.00076 [0.00071 to 0.00085] | 0.00076 [0.00064 to 0.00094] | 0.00071 [0.00067 to 0.00086] | 0.0008 [0.000755 to 0.000945] | 0.000735 [0.00068 to 0.00096] |
  Creatinine (g/dL)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 57 - 71 | 0.00076 [0.00071 to 0.00081] | 0.00076 [0.00061 to 0.00086] |  |  |  |
  Creatinine (g/dL)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Creatinine (g/dL)- Day 99 - 113 |  |  | 0.00078 [0.00067 to 0.00089] |  |  |
  Creatinine (g/dL)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Creatinine (g/dL)- Day 127 - 141 | 0.00074 [0.00063 to 0.00079] | 0.000735 [0.00063 to 0.00084] |  | 0.00081 [0.00073 to 0.00091] |  |
  Creatinine (g/dL)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  Creatinine (g/dL)- Day 169 - 183 | 0.00073 [0.00064 to 0.00077] | 0.0008 [0.000645 to 0.000905] | 0.000765 [0.00072 to 0.00082] |  |  |
  Creatinine (g/dL)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Creatinine (g/dL)- Day 252 - 267 | 0.000715 [0.000625 to 0.000775] | 0.00072 [0.00068 to 0.00085] |  |  | 0.00077 [0.00073 to 0.000875] |
  Creatinine (g/dL)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Creatinine (g/dL)- Day 442 - 456 |  |  | 0.00082 [0.00074 to 0.00096] |  |  |

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC)
Description: Chemistry and Hematology Laboratory Measures - lymphocyte count (1000/mm3), neutrophil count (1000/mm3), platelets (1000/mm3), white blood cells (WBC) (1000/mm3)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: 1000/mm3
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1
1000/mm3
  WBC (1000/cubic mm)- Screening | 6.37 [5.6 to 8.48] | 7.14 [6.24 to 8.39] | 8.31 [6.35 to 8.5] | 5.85 [4.45 to 7.15] | 6.45 [5.4 to 7.7] | 9.02 [9.02 to 9.02]
  WBC (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  WBC (1000/cubic mm)- Day 1 - 15 | 5.9 [5.31 to 7.98] | 5.86 [4.91 to 7.28] | 6.53 [5.91 to 7.51] | 5.2 [4.2 to 6.45] | 6.35 [5.4 to 7.1] |
  WBC (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 57 - 71 | 6.21 [4.95 to 7.11] | 7.26 [5.4 to 8.33] |  |  |  |
  WBC (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 99 - 113 |  |  | 5.5 [4.72 to 7.91] |  |  |
  WBC (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  WBC (1000/cubic mm)- Day 127 - 141 | 6.395 [5.01 to 8.33] | 6.475 [5.065 to 7.035] |  | 5.5 [4.4 to 6.6] |  |
  WBC (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 169 - 183 | 5.83 [4.34 to 6.665] | 6.2 [5.25 to 8] | 6.5 [5.31 to 7.11] |  |  |
  WBC (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  WBC (1000/cubic mm)- Day 252 - 267 | 6.21 [4.885 to 7.82] | 6.92 [5.14 to 7.81] |  |  | 6.45 [5.6 to 7.1] |
  WBC (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 442 - 456 |  |  | 5.67 [4.99 to 6.38] |  |  |
  Neutrophils (1000/cubic mm)- Screening | 3.709 [2.996 to 5.357] | 4.185 [3.14 to 4.76] | 4.958 [4 to 5.32] | 3.494 [2.1795 to 4.215] | 3.4345 [2.604 to 5.028] | 6.747 [6.747 to 6.747]
  Neutrophils (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Neutrophils (1000/cubic mm)- Day 1 - 15 | 3.336 [2.51 to 5.05] | 3.54 [2.468 to 4.16] | 3.853 [3.377 to 5.43] | 3.124 [2.2245 to 3.7045] | 3.733 [3.089 to 3.919] |
  Neutrophils (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 57 - 71 | 3.3 [2.42 to 5.137] | 4 [2.984 to 4.615] |  |  |  |
  Neutrophils (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 99 - 113 |  |  | 3.27 [2.57 to 4.516] |  |  |
  Neutrophils (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 127 - 141 | 3.8025 [2.875 to 5.0905] | 3.4375 [2.5165 to 4.4505] |  | 3.26 [2.494 to 3.907] |  |
  Neutrophils (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 169 - 183 | 3.63 [2.2105 to 4.2] | 3.14 [2.796 to 4.41] | 3.775 [3.159 to 4.264] |  |  |
  Neutrophils (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Neutrophils (1000/cubic mm)- Day 252 - 267 | 4.0245 [2.638 to 5.07] | 3.599 [2.66 to 5.05] |  |  | 3.301 [2.8055 to 3.9125] |
  Neutrophils (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 442 - 456 |  |  | 3.02 [2.51 to 3.42] |  |  |
  Lymphocytes (1000/cubic mm)- Screening | 2.033 [1.793 to 2.32] | 2.198 [1.98 to 2.69] | 2.255 [1.81 to 3.22] | 1.875 [1.37 to 2.284] | 2.161 [1.62 to 2.85] | 1.741 [1.741 to 1.741]
  Lymphocytes (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Lymphocytes (1000/cubic mm)- Day 1 - 15 | 1.93 [1.561 to 2.42] | 1.872 [1.562 to 2.48] | 2.21 [1.65 to 2.589] | 1.68 [1.39 to 1.9645] | 2.0345 [1.86 to 2.347] |
  Lymphocytes (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 57 - 71 | 1.7 [1.57 to 2.29] | 2.27 [1.58 to 2.62] |  |  |  |
  Lymphocytes (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 99 - 113 |  |  | 1.743 [1.54 to 2.079] |  |  |
  Lymphocytes (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 127 - 141 | 1.843 [1.4225 to 2.334] | 2.09 [1.5 to 2.58] |  | 1.72 [1.33 to 2.17] |  |
  Lymphocytes (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 169 - 183 | 1.7685 [1.46 to 2.0765] | 1.966 [1.58 to 2.49] | 1.7765 [1.608 to 2.14] |  |  |
  Lymphocytes (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Lymphocytes (1000/cubic mm)- Day 252 - 267 | 1.8045 [1.465 to 2.085] | 1.95 [1.576 to 2.45] |  |  | 2.251 [2.0645 to 2.342] |
  Lymphocytes (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 442 - 456 |  |  | 2.156 [1.52 to 2.82] |  |  |
  Platelets (1000/cubic mm)- Screening | 256 [226 to 292] | 275 [203 to 314] | 281 [238 to 374] | 258 [229.5 to 301] | 270.5 [245 to 314] | 334 [334 to 334]
  Platelets (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Platelets (1000/cubic mm)- Day 1 - 15 | 255 [225 to 291] | 274 [203 to 305] | 285 [251 to 366] | 258.5 [213 to 302] | 278 [212 to 312] |
  Platelets (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 57 - 71 | 247 [210 to 279] | 285 [214 to 319] |  |  |  |
  Platelets (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 99 - 113 |  |  | 290 [265 to 305] |  |  |
  Platelets (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Platelets (1000/cubic mm)- Day 127 - 141 | 258 [228 to 323.5] | 294 [220 to 312] |  | 274 [218 to 310] |  |
  Platelets (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 169 - 183 | 249 [217 to 274] | 261 [197 to 302] | 278 [260 to 415] |  |  |
  Platelets (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 20 | 0 | 0 | 8 | 0
  Platelets (1000/cubic mm)- Day 252 - 267 | 253 [221.5 to 276] | 266.5 [224.5 to 308.5] |  |  | 259.5 [194 to 325.5] |
  Platelets (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 442 - 456 |  |  | 269 [229 to 336] |  |  |

6. Primary Outcome: Number of Participants With Chemistry and Hematology Laboratory Measures - Counts of Lab Grade > 1
Description: Number of Participants with Chemistry and Hematology Laboratory Measures - Counts of Lab Grade > 1 for alkaline phosphate (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC).
Time Frame: as for outcome 3
Population: Visit schedule is not the same for each treatment group. For visits not on the schedule, number analyzed is 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1
Participants
  WBC (1000/cubic mm)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  WBC (1000/cubic mm)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  WBC (1000/cubic mm)- Day 127 - 141 | 0 | 0 | 0 | 1 | 0 | 0
  WBC (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  WBC (1000/cubic mm)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  WBC (1000/cubic mm)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Neutrophils (1000/cubic mm)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 127 - 141 | 0 | 0 | 0 | 1 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Neutrophils (1000/cubic mm)- Day 252 - 267 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Hemoglobin (g/dL)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Hemoglobin (g/dL)- Day 127 - 141 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Hemoglobin (g/dL)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Lymphocytes (1000/cubic mm)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 127 - 141 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Lymphocytes (1000/cubic mm)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Platelets (1000/cubic mm)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Platelets (1000/cubic mm)- Day 127 - 141 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets (1000/cubic mm)- Day 169 - 183: number analyzed (Participants) | 20 | 19 | 6 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 252 - 267: number analyzed (Participants) | 20 | 20 | 0 | 0 | 8 | 0
  Platelets (1000/cubic mm)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Platelets (1000/cubic mm)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  ALT (SGPT) (U/L)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  ALT (SGPT) (U/L)- Day 127 - 141 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 1 | 0 | 8 | 0
  ALT (SGPT) (U/L)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  AST (U/L)- Day 1 - 15 | 0 | 0 | 0 | 1 | 0 | 0
  AST (U/L)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  AST (U/L)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  AST (U/L)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  AST (U/L)- Day 127 - 141 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  AST (U/L)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  AST (U/L)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  AST (U/L)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  AST (U/L)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Alkaline Phosphatase (U/L)- Day 1 - 15 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 57 - 71 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 127 - 141 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 169 - 183 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Alkaline Phosphatase (U/L)- Day 252 - 267 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- DayScreening | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 1 - 15: number analyzed (Participants) | 21 | 23 | 7 | 16 | 10 | 0
  Creatinine (g/dL)- Day 1 - 15 | 1 | 1 | 1 | 0 | 0 | 0
  Creatinine (g/dL)- Day 57 - 71: number analyzed (Participants) | 21 | 21 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 57 - 71 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 99 - 113: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 0
  Creatinine (g/dL)- Day 99 - 113 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 127 - 141: number analyzed (Participants) | 20 | 20 | 0 | 15 | 0 | 0
  Creatinine (g/dL)- Day 127 - 141 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 169 - 183: number analyzed (Participants) | 20 | 20 | 6 | 0 | 0 | 0
  Creatinine (g/dL)- Day 169 - 183 | 0 | 3 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 252 - 267: number analyzed (Participants) | 20 | 21 | 0 | 0 | 8 | 0
  Creatinine (g/dL)- Day 252 - 267 | 1 | 1 | 0 | 0 | 0 | 0
  Creatinine (g/dL)- Day 442 - 456: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Creatinine (g/dL)- Day 442 - 456 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: For participants reporting multiple AEs over the time frame, the maximum severity is counted
Time Frame: Measured through participant's last study visit, at 6 months to 1 1/2 years after study entry (depending on which group participants are in)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1
Participants
  Mild | 5 | 3 | 0 | 2 | 1 | 1
  Moderate | 16 | 11 | 6 | 5 | 1 | 0
  Severe | 1 | 4 | 1 | 0 | 1 | 0
  Potentially life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  No AE reported | 1 | 5 | 0 | 9 | 7 | 0

8. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: For participants reporting multiple AEs over the time frame, the maximum severity is counted
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10 | 1
Participants
  SAE | 0 | 1 | 1 | 0 | 1 | 0
  No SAE reported | 23 | 22 | 6 | 16 | 9 | 1

9. Primary Outcome: Rates of Participant Discontinuation
Description: Tabulated by reason for discontinuation and treatment arm
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine
Number analyzed (Participants) | 23 | 23 | 7 | 16 | 10
Participants
  Coenrolled with an investigational agent | 1 | 0 | 0 | 0 | 0
  Terminated to donate bone marrow | 0 | 1 | 0 | 0 | 0
  Refused study product administration | 1 | 0 | 0 | 0 | 0
  Clinical event (not reacto, HIV, death) | 1 | 0 | 1 | 0 | 0
  Unable to contact participant for visits | 1 | 0 | 0 | 0 | 0
  Did not discontinue SPA | 19 | 22 | 6 | 16 | 10

10. Primary Outcome: Unnormalized Serum Concentration of VRC01 Out to Month 6 After the Last Infusion (for Groups 1, 2, and 4)
Description: Outcome measure will not be ready before the anticipated reporting date. VRC01/LS levels were measured by Singulex assay. VRC01/LS levels of study samples are calibrated via the respective standard curve on each assay plate. A five-parameter logistic (5PL) model is used to fit the standard curve data using the nCal package in R. Outcome measure is the estimated concentration of VRC01/VRC01LS.
Time Frame: Measured through 6 months after the last infusion
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 4: Vaccine
Number analyzed (Participants) | 23 | 23 | 16
µg/mL
  Serum-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Serum-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Serum-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Serum-Female-Visit 2 | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] |
  Serum-Male-Visit 2: number analyzed (Participants) | 10 | 10 | 0
  Serum-Male-Visit 2 | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] |
  Serum-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 8
  Serum-Female-Visit 3 |  |  | 0.05 [0.02 to 0.08]
  Serum-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 8
  Serum-Male-Visit 3 |  |  | 0.05 [0.02 to 0.13]
  Serum-Female-Visit 4: number analyzed (Participants) | 12 | 13 | 8
  Serum-Female-Visit 4 | 72.42 [62.99 to 99.58] | 215.65 [172.82 to 271.26] | 194.99 [177.75 to 215.86]
  Serum-Male-Visit 4: number analyzed (Participants) | 9 | 10 | 8
  Serum-Male-Visit 4 | 64.83 [48.7 to 129.28] | 185.55 [140.18 to 211.36] | 240.46 [220.3 to 335.77]
  Serum-Female-Visit 5: number analyzed (Participants) | 13 | 12 | 5
  Serum-Female-Visit 5 | 19.77 [14.53 to 25.6] | 49.27 [41.83 to 62.52] | 72.31 [71.59 to 73.77]
  Serum-Male-Visit 5: number analyzed (Participants) | 10 | 10 | 6
  Serum-Male-Visit 5 | 19.57 [10.11 to 24.03] | 54.09 [40.84 to 58.16] | 60.48 [53.49 to 74.24]
  Serum-Female-Visit 7: number analyzed (Participants) | 12 | 11 | 8
  Serum-Female-Visit 7 | 50.95 [42.03 to 82.81] | 202.99 [153.76 to 271.53] | 29.72 [19.91 to 36.55]
  Serum-Male-Visit 7: number analyzed (Participants) | 9 | 9 | 7
  Serum-Male-Visit 7 | 62.08 [52.76 to 105.56] | 274.67 [227.19 to 364.53] | 20.99 [15.45 to 38.65]
  Serum-Female-Visit 9: number analyzed (Participants) | 12 | 11 | 8
  Serum-Female-Visit 9 | 13.48 [7.85 to 18.73] | 54.76 [43.67 to 63.84] | 8.51 [6.55 to 12.15]
  Serum-Male-Visit 9: number analyzed (Participants) | 8 | 9 | 7
  Serum-Male-Visit 9 | 14.84 [13.27 to 17.46] | 49.05 [46.68 to 53.2] | 5.81 [4.14 to 16.84]
  Serum-Female-Visit 12: number analyzed (Participants) | 8 | 10 | 7
  Serum-Female-Visit 12 | 29.11 [22.83 to 36.53] | 112.28 [94.48 to 128] | 1.65 [1.3 to 2.72]
  Serum-Male-Visit 12: number analyzed (Participants) | 7 | 10 | 7
  Serum-Male-Visit 12 | 36.48 [28.65 to 51.21] | 104.97 [94.57 to 116.37] | 1.71 [1.05 to 4.85]
  Serum-Female-Visit 14: number analyzed (Participants) | 13 | 10 | 7
  Serum-Female-Visit 14 | 81.92 [63.44 to 104.76] | 174.79 [132.71 to 226.69] | 0.66 [0.55 to 0.84]
  Serum-Male-Visit 14: number analyzed (Participants) | 7 | 9 | 7
  Serum-Male-Visit 14 | 72.35 [59.34 to 150.89] | 228.43 [191.91 to 264.03] | 0.67 [0.48 to 1.06]
  Serum-Female-Visit 15: number analyzed (Participants) | 12 | 10 | 0
  Serum-Female-Visit 15 | 9.6 [8.64 to 16.55] | 26.85 [21.48 to 32.15] |
  Serum-Male-Visit 15: number analyzed (Participants) | 6 | 9 | 0
  Serum-Male-Visit 15 | 11.5 [8.73 to 51.29] | 62.81 [41.08 to 79.96] |
  Serum-Female-Visit 16: number analyzed (Participants) | 11 | 11 | 0
  Serum-Female-Visit 16 | 1.25 [0.64 to 1.96] | 3.03 [1.7 to 7.35] |
  Serum-Male-Visit 16: number analyzed (Participants) | 6 | 10 | 0
  Serum-Male-Visit 16 | 1.12 [0.73 to 4.82] | 6.85 [3.02 to 18.29] |
  Serum-Female-Visit 17: number analyzed (Participants) | 8 | 10 | 0
  Serum-Female-Visit 17 | 0.02 [0.02 to 0.1] | 0.11 [0.08 to 0.55] |
  Serum-Male-Visit 17: number analyzed (Participants) | 6 | 8 | 0
  Serum-Male-Visit 17 | 0.03 [0.02 to 0.17] | 0.15 [0.05 to 0.43] |

11. Primary Outcome: IgG-normalized Serum Concentration of VRC01 Out to Month 6 After the Last Infusion (for Groups 1, 2, and 4)
Description: Outcome measure will not be ready before the anticipated reporting date. VRC01/LS levels were measured by Singulex assay. VRC01/LS levels and total IgG levels of study samples are calibrated via the respective standard curve on each assay plate. A five-parameter logistic (5PL) model is used to fit the standard curve data using the nCal package in R. Outcome measure is the IgG-normalized VRC01/VRC01LS levels performed by dividing VRC01/LS levels (pg/mL) by the total IgG concentrations (ng/mL)
Time Frame: Measured through 6 months after the last infusion
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng IgG
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 4: Vaccine
Number analyzed (Participants) | 23 | 23 | 16
pg mAb/ng IgG
  Serum-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Serum-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Serum-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Serum-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Serum-Male-Visit 2: number analyzed (Participants) | 10 | 10 | 0
  Serum-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Serum-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 8
  Serum-Female-Visit 3 |  |  | 0 [0 to 0.01]
  Serum-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 8
  Serum-Male-Visit 3 |  |  | 0.01 [0 to 0.01]
  Serum-Female-Visit 4: number analyzed (Participants) | 12 | 13 | 8
  Serum-Female-Visit 4 | 6.28 [4.98 to 7.32] | 13.82 [11.41 to 23.35] | 17.02 [16.1 to 25.71]
  Serum-Male-Visit 4: number analyzed (Participants) | 9 | 10 | 8
  Serum-Male-Visit 4 | 6.8 [3.61 to 10.16] | 12.94 [8.1 to 16.54] | 22.1 [17.5 to 27.14]
  Serum-Female-Visit 5: number analyzed (Participants) | 13 | 12 | 5
  Serum-Female-Visit 5 | 1.54 [0.73 to 2.68] | 4 [2.52 to 5.09] | 7.09 [4.28 to 9.57]
  Serum-Male-Visit 5: number analyzed (Participants) | 10 | 10 | 6
  Serum-Male-Visit 5 | 1.44 [0.69 to 2.89] | 3.59 [2.49 to 5.02] | 5.48 [3.4 to 7.25]
  Serum-Female-Visit 7: number analyzed (Participants) | 12 | 11 | 8
  Serum-Female-Visit 7 | 4.26 [2.78 to 7.3] | 19.67 [11.04 to 23.09] | 2.31 [1.84 to 3.48]
  Serum-Male-Visit 7: number analyzed (Participants) | 9 | 9 | 7
  Serum-Male-Visit 7 | 5.75 [3.28 to 7.04] | 23.75 [19.2 to 24.5] | 1.62 [1.07 to 2.32]
  Serum-Female-Visit 9: number analyzed (Participants) | 12 | 11 | 8
  Serum-Female-Visit 9 | 0.9 [0.63 to 1.68] | 3.61 [3.26 to 4.49] | 0.79 [0.54 to 1.17]
  Serum-Male-Visit 9: number analyzed (Participants) | 8 | 9 | 7
  Serum-Male-Visit 9 | 1 [0.83 to 1.74] | 3.55 [2.92 to 5.13] | 0.41 [0.31 to 1.32]
  Serum-Female-Visit 12: number analyzed (Participants) | 8 | 10 | 7
  Serum-Female-Visit 12 | 1.94 [1.26 to 2.76] | 8.41 [6.4 to 11.49] | 0.15 [0.11 to 0.25]
  Serum-Male-Visit 12: number analyzed (Participants) | 7 | 10 | 7
  Serum-Male-Visit 12 | 3.07 [1.49 to 4.68] | 7.49 [5.81 to 9.33] | 0.13 [0.07 to 0.34]
  Serum-Female-Visit 14: number analyzed (Participants) | 13 | 10 | 7
  Serum-Female-Visit 14 | 6.55 [4.24 to 10.13] | 13.11 [8.17 to 19.83] | 0.06 [0.05 to 0.07]
  Serum-Male-Visit 14: number analyzed (Participants) | 7 | 9 | 7
  Serum-Male-Visit 14 | 7.13 [5.29 to 13.1] | 21.79 [11.23 to 24.13] | 0.06 [0.03 to 0.08]
  Serum-Female-Visit 15: number analyzed (Participants) | 12 | 10 | 0
  Serum-Female-Visit 15 | 0.78 [0.63 to 1.43] | 1.88 [1.11 to 3.41] |
  Serum-Male-Visit 15: number analyzed (Participants) | 6 | 9 | 0
  Serum-Male-Visit 15 | 0.84 [0.57 to 5.41] | 3.38 [2.91 to 5.56] |
  Serum-Female-Visit 16: number analyzed (Participants) | 11 | 11 | 0
  Serum-Female-Visit 16 | 0.09 [0.04 to 0.12] | 0.17 [0.14 to 0.74] |
  Serum-Male-Visit 16: number analyzed (Participants) | 6 | 10 | 0
  Serum-Male-Visit 16 | 0.08 [0.05 to 0.48] | 0.39 [0.16 to 1.72] |
  Serum-Female-Visit 17: number analyzed (Participants) | 8 | 10 | 0
  Serum-Female-Visit 17 | 0 [0 to 0.01] | 0.01 [0 to 0.05] |
  Serum-Male-Visit 17: number analyzed (Participants) | 6 | 8 | 0
  Serum-Male-Visit 17 | 0 [0 to 0.01] | 0.01 [0 to 0.03] |

12. Primary Outcome: Protein-normalized Serum Concentration of VRC01 Out to Month 6 After the Last Infusion (for Groups 1, 2, and 4)
Description: Outcome measure will not be ready before the anticipated reporting date. VRC01/LS levels were measured by Singulex assay. VRC01/LS levels and total protein levels of study samples are calibrated via the respective standard curve on each assay plate. A five-parameter logistic (5PL) model is used to fit the standard curve data using the nCal package in R. Outcome measure is the protein-normalized VRC01/VRC01LS levels performed by dividing VRC01/LS levels (pg/mL) by the total protein concentrations (ng/mL)
Time Frame: Measured through 6 months after the last infusion
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng total protein
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 4: Vaccine
Number analyzed (Participants) | 23 | 23 | 16
pg mAb/ng total protein
  Serum-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Serum-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Serum-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Serum-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Serum-Male-Visit 2: number analyzed (Participants) | 10 | 10 | 0
  Serum-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Serum-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 8
  Serum-Female-Visit 3 |  |  | 0 [0 to 0]
  Serum-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 8
  Serum-Male-Visit 3 |  |  | 0 [0 to 0]
  Serum-Female-Visit 4: number analyzed (Participants) | 12 | 13 | 8
  Serum-Female-Visit 4 | 0.87 [0.7 to 1.01] | 2.5 [1.89 to 3.15] | 2.39 [1.89 to 2.79]
  Serum-Male-Visit 4: number analyzed (Participants) | 9 | 10 | 8
  Serum-Male-Visit 4 | 0.78 [0.48 to 1.64] | 2.04 [1.74 to 2.45] | 2.77 [2.29 to 3.7]
  Serum-Female-Visit 5: number analyzed (Participants) | 13 | 12 | 5
  Serum-Female-Visit 5 | 0.21 [0.17 to 0.28] | 0.6 [0.52 to 0.76] | 0.88 [0.8 to 0.91]
  Serum-Male-Visit 5: number analyzed (Participants) | 10 | 10 | 6
  Serum-Male-Visit 5 | 0.21 [0.12 to 0.27] | 0.65 [0.5 to 0.7] | 0.63 [0.56 to 0.84]
  Serum-Female-Visit 7: number analyzed (Participants) | 12 | 11 | 8
  Serum-Female-Visit 7 | 0.66 [0.47 to 0.92] | 2.34 [1.76 to 3.19] | 0.33 [0.22 to 0.4]
  Serum-Male-Visit 7: number analyzed (Participants) | 9 | 9 | 7
  Serum-Male-Visit 7 | 0.67 [0.63 to 1.3] | 3.66 [2.49 to 3.83] | 0.19 [0.17 to 0.43]
  Serum-Female-Visit 9: number analyzed (Participants) | 12 | 11 | 8
  Serum-Female-Visit 9 | 0.16 [0.1 to 0.21] | 0.68 [0.45 to 0.74] | 0.1 [0.08 to 0.15]
  Serum-Male-Visit 9: number analyzed (Participants) | 8 | 9 | 7
  Serum-Male-Visit 9 | 0.18 [0.14 to 0.21] | 0.6 [0.52 to 0.61] | 0.06 [0.05 to 0.23]
  Serum-Female-Visit 12: number analyzed (Participants) | 8 | 10 | 7
  Serum-Female-Visit 12 | 0.35 [0.26 to 0.44] | 1.22 [1.1 to 1.29] | 0.02 [0.02 to 0.03]
  Serum-Male-Visit 12: number analyzed (Participants) | 7 | 10 | 7
  Serum-Male-Visit 12 | 0.39 [0.3 to 0.56] | 1.22 [1.12 to 1.34] | 0.02 [0.01 to 0.06]
  Serum-Female-Visit 14: number analyzed (Participants) | 13 | 10 | 7
  Serum-Female-Visit 14 | 0.9 [0.73 to 1.2] | 2.07 [1.59 to 2.48] | 0.01 [0.01 to 0.01]
  Serum-Male-Visit 14: number analyzed (Participants) | 7 | 9 | 7
  Serum-Male-Visit 14 | 0.84 [0.56 to 1.62] | 2.59 [2.18 to 2.8] | 0.01 [0.01 to 0.01]
  Serum-Female-Visit 15: number analyzed (Participants) | 12 | 10 | 0
  Serum-Female-Visit 15 | 0.1 [0.1 to 0.17] | 0.32 [0.26 to 0.41] |
  Serum-Male-Visit 15: number analyzed (Participants) | 6 | 9 | 0
  Serum-Male-Visit 15 | 0.15 [0.1 to 0.54] | 0.69 [0.4 to 0.71] |
  Serum-Female-Visit 16: number analyzed (Participants) | 11 | 11 | 0
  Serum-Female-Visit 16 | 0.02 [0.01 to 0.02] | 0.03 [0.02 to 0.1] |
  Serum-Male-Visit 16: number analyzed (Participants) | 6 | 10 | 0
  Serum-Male-Visit 16 | 0.01 [0.01 to 0.06] | 0.07 [0.03 to 0.2] |
  Serum-Female-Visit 17: number analyzed (Participants) | 8 | 10 | 0
  Serum-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0.01] |
  Serum-Male-Visit 17: number analyzed (Participants) | 6 | 8 | 0
  Serum-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |

13. Primary Outcome: Unnormalized Levels of VRC01 in Genital and Rectal Secretions, as Well as Cervical, Vaginal, and Rectal Tissues (for Groups 1, 2, and 4)
Description: as for outcome 10
Time Frame: Measured through 6 months after the last infusion
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 4: Vaccine
Number analyzed (Participants) | 23 | 23 | 16
µg/mL
  Cervical Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Cervical Biopsy Lysate-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Cervical Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Cervical Biopsy Lysate-Female-Visit 4 |  |  | 0.9 [0.86 to 1]
  Cervical Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 5
  Cervical Biopsy Lysate-Female-Visit 5 |  |  | 0.26 [0.17 to 0.29]
  Cervical Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 8
  Cervical Biopsy Lysate-Female-Visit 9 |  |  | 0.03 [0.03 to 0.04]
  Cervical Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Cervical Biopsy Lysate-Female-Visit 12 |  |  | 0.01 [0.01 to 0.03]
  Cervical Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 9 | 9 | 7
  Cervical Biopsy Lysate-Female-Visit 14 | 0.28 [0.22 to 0.39] | 0.91 [0.77 to 1.08] | 0.01 [0.01 to 0.02]
  Cervical Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 9 | 9 | 0
  Cervical Biopsy Lysate-Female-Visit 15 | 0.06 [0.03 to 0.06] | 0.17 [0.08 to 0.19] |
  Cervical Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 7 | 7 | 0
  Cervical Biopsy Lysate-Female-Visit 16 | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.03] |
  Cervical Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 6 | 7 | 0
  Cervical Biopsy Lysate-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Cervical Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 7 | 5 | 0
  Rectal Biopsy Lysate-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 9 | 10 | 0
  Rectal Biopsy Lysate-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Rectal Biopsy Lysate-Male-Visit 4 |  |  | 0.33 [0.24 to 0.43]
  Rectal Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 6
  Rectal Biopsy Lysate-Male-Visit 5 |  |  | 0.09 [0.07 to 0.15]
  Rectal Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 7
  Rectal Biopsy Lysate-Male-Visit 9 |  |  | 0.01 [0 to 0.01]
  Rectal Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Rectal Biopsy Lysate-Male-Visit 12 |  |  | 0 [0 to 0.01]
  Rectal Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 6 | 2 | 0
  Rectal Biopsy Lysate-Female-Visit 14 | 0.1 [0.09 to 0.12] | 0.16 [0.13 to 0.18] |
  Rectal Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 5 | 8 | 7
  Rectal Biopsy Lysate-Male-Visit 14 | 0.06 [0.03 to 0.11] | 0.23 [0.19 to 0.32] | 0 [0 to 0]
  Rectal Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 6 | 5 | 0
  Rectal Biopsy Lysate-Female-Visit 15 | 0.02 [0.01 to 0.04] | 0.04 [0.02 to 0.05] |
  Rectal Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 6 | 8 | 0
  Rectal Biopsy Lysate-Male-Visit 15 | 0.02 [0.01 to 0.02] | 0.06 [0.05 to 0.11] |
  Rectal Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 4 | 4 | 0
  Rectal Biopsy Lysate-Female-Visit 16 | 0 [0 to 0.01] | 0.01 [0 to 0.01] |
  Rectal Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 6 | 9 | 0
  Rectal Biopsy Lysate-Male-Visit 16 | 0 [0 to 0] | 0.01 [0 to 0.01] |
  Rectal Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 1 | 4 | 0
  Rectal Biopsy Lysate-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 4 | 9 | 0
  Rectal Biopsy Lysate-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 7
  Rectal Secretions-Male-Visit 1 |  |  | 0 [0 to 0]
  Rectal Secretions-Female-Visit 2: number analyzed (Participants) | 7 | 6 | 0
  Rectal Secretions-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 2: number analyzed (Participants) | 7 | 10 | 0
  Rectal Secretions-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Female-Visit 4: number analyzed (Participants) | 7 | 6 | 0
  Rectal Secretions-Female-Visit 4 | 0 [0 to 0.01] | 0 [0 to 0.01] |
  Rectal Secretions-Male-Visit 4: number analyzed (Participants) | 7 | 8 | 6
  Rectal Secretions-Male-Visit 4 | 0 [0 to 0.01] | 0.02 [0 to 0.09] | 0.01 [0.01 to 0.01]
  Rectal Secretions-Female-Visit 5: number analyzed (Participants) | 6 | 5 | 0
  Rectal Secretions-Female-Visit 5 | 0 [0 to 0] | 0 [0 to 0.05] |
  Rectal Secretions-Male-Visit 5: number analyzed (Participants) | 7 | 10 | 6
  Rectal Secretions-Male-Visit 5 | 0 [0 to 0] | 0 [0 to 0.01] | 0 [0 to 0.01]
  Rectal Secretions-Female-Visit 7: number analyzed (Participants) | 6 | 5 | 0
  Rectal Secretions-Female-Visit 7 | 0 [0 to 0] | 0.01 [0 to 0.01] |
  Rectal Secretions-Male-Visit 7: number analyzed (Participants) | 7 | 6 | 6
  Rectal Secretions-Male-Visit 7 | 0.01 [0 to 0.01] | 0.02 [0.01 to 0.11] | 0 [0 to 0.01]
  Rectal Secretions-Female-Visit 9: number analyzed (Participants) | 5 | 5 | 0
  Rectal Secretions-Female-Visit 9 | 0 [0 to 0] | 0.01 [0 to 0.01] |
  Rectal Secretions-Male-Visit 9: number analyzed (Participants) | 4 | 7 | 7
  Rectal Secretions-Male-Visit 9 | 0 [0 to 0] | 0 [0 to 0.04] | 0 [0 to 0]
  Rectal Secretions-Female-Visit 12: number analyzed (Participants) | 3 | 4 | 0
  Rectal Secretions-Female-Visit 12 | 0 [0 to 0] | 0 [0 to 0.01] |
  Rectal Secretions-Male-Visit 12: number analyzed (Participants) | 4 | 7 | 6
  Rectal Secretions-Male-Visit 12 | 0 [0 to 0.01] | 0 [0 to 0.01] | 0 [0 to 0]
  Rectal Secretions-Female-Visit 14: number analyzed (Participants) | 7 | 3 | 0
  Rectal Secretions-Female-Visit 14 | 0 [0 to 0.02] | 0 [0 to 0.01] |
  Rectal Secretions-Male-Visit 14: number analyzed (Participants) | 5 | 8 | 6
  Rectal Secretions-Male-Visit 14 | 0 [0 to 0.04] | 0 [0 to 0.03] | 0 [0 to 0]
  Rectal Secretions-Female-Visit 15: number analyzed (Participants) | 5 | 5 | 0
  Rectal Secretions-Female-Visit 15 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 15: number analyzed (Participants) | 4 | 5 | 0
  Rectal Secretions-Male-Visit 15 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Female-Visit 16: number analyzed (Participants) | 2 | 4 | 0
  Rectal Secretions-Female-Visit 16 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 16: number analyzed (Participants) | 4 | 7 | 0
  Rectal Secretions-Male-Visit 16 | 0 [0 to 0] | 0 [0 to 0.01] |
  Rectal Secretions-Female-Visit 17: number analyzed (Participants) | 1 | 3 | 0
  Rectal Secretions-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 17: number analyzed (Participants) | 4 | 7 | 0
  Rectal Secretions-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Semen-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 8
  Semen-Male-Visit 1 |  |  | 0 [0 to 0]
  Semen-Female-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 2: number analyzed (Participants) | 10 | 9 | 0
  Semen-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Semen-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Semen-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 4: number analyzed (Participants) | 8 | 10 | 8
  Semen-Male-Visit 4 | 0.15 [0.08 to 0.2] | 0.43 [0.37 to 0.56] | 0.49 [0.3 to 0.58]
  Semen-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 5: number analyzed (Participants) | 10 | 10 | 6
  Semen-Male-Visit 5 | 0.05 [0.02 to 0.06] | 0.14 [0.09 to 0.2] | 0.16 [0.14 to 0.26]
  Semen-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 7: number analyzed (Participants) | 9 | 9 | 7
  Semen-Male-Visit 7 | 0.14 [0.11 to 0.19] | 0.46 [0.34 to 0.62] | 0.05 [0.04 to 0.09]
  Semen-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 9: number analyzed (Participants) | 8 | 9 | 7
  Semen-Male-Visit 9 | 0.04 [0.03 to 0.07] | 0.17 [0.12 to 0.19] | 0.02 [0.01 to 0.03]
  Semen-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 12: number analyzed (Participants) | 7 | 10 | 7
  Semen-Male-Visit 12 | 0.12 [0.1 to 0.15] | 0.32 [0.25 to 0.34] | 0 [0 to 0.01]
  Semen-Female-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 14: number analyzed (Participants) | 7 | 9 | 7
  Semen-Male-Visit 14 | 0.13 [0.1 to 0.17] | 0.42 [0.36 to 0.87] | 0 [0 to 0]
  Semen-Female-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 15: number analyzed (Participants) | 6 | 9 | 0
  Semen-Male-Visit 15 | 0.04 [0.02 to 0.06] | 0.12 [0.07 to 0.2] |
  Semen-Female-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 16: number analyzed (Participants) | 6 | 10 | 0
  Semen-Male-Visit 16 | 0.01 [0 to 0.02] | 0.01 [0.01 to 0.02] |
  Semen-Female-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 17: number analyzed (Participants) | 6 | 9 | 0
  Semen-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Softcup Fluid-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 5
  Softcup Fluid-Female-Visit 1 |  |  | 0.02 [0.01 to 0.02]
  Softcup Fluid-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 2: number analyzed (Participants) | 6 | 7 | 0
  Softcup Fluid-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0.01] |
  Softcup Fluid-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 4: number analyzed (Participants) | 4 | 2 | 5
  Softcup Fluid-Female-Visit 4 | 0.28 [0.23 to 0.5] | 0.67 [0.59 to 0.75] | 0.93 [0.8 to 1.27]
  Softcup Fluid-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 5: number analyzed (Participants) | 4 | 4 | 2
  Softcup Fluid-Female-Visit 5 | 0.04 [0.02 to 0.07] | 0.16 [0.1 to 0.33] | 0.2 [0.18 to 0.21]
  Softcup Fluid-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 7: number analyzed (Participants) | 7 | 6 | 5
  Softcup Fluid-Female-Visit 7 | 0.29 [0.17 to 0.31] | 0.97 [0.73 to 1.43] | 0.08 [0.03 to 0.14]
  Softcup Fluid-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 9: number analyzed (Participants) | 7 | 6 | 4
  Softcup Fluid-Female-Visit 9 | 0.04 [0.04 to 0.08] | 0.24 [0.21 to 0.27] | 0.06 [0.04 to 0.08]
  Softcup Fluid-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 12: number analyzed (Participants) | 2 | 4 | 5
  Softcup Fluid-Female-Visit 12 | 0.43 [0.34 to 0.52] | 0.71 [0.49 to 1.16] | 0.01 [0.01 to 0.01]
  Softcup Fluid-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 14: number analyzed (Participants) | 6 | 6 | 3
  Softcup Fluid-Female-Visit 14 | 0.33 [0.26 to 0.4] | 0.6 [0.28 to 0.91] | 0.01 [0 to 0.01]
  Softcup Fluid-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 15: number analyzed (Participants) | 7 | 6 | 0
  Softcup Fluid-Female-Visit 15 | 0.09 [0.04 to 0.11] | 0.09 [0.03 to 0.17] |
  Softcup Fluid-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 16: number analyzed (Participants) | 4 | 4 | 0
  Softcup Fluid-Female-Visit 16 | 0.01 [0.01 to 0.01] | 0.04 [0.01 to 0.14] |
  Softcup Fluid-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 17: number analyzed (Participants) | 4 | 5 | 0
  Softcup Fluid-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0.01] |
  Softcup Fluid-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Vaginal Biopsy Lysate-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Vaginal Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Vaginal Biopsy Lysate-Female-Visit 4 |  |  | 0.7 [0.55 to 1.4]
  Vaginal Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 5
  Vaginal Biopsy Lysate-Female-Visit 5 |  |  | 0.29 [0.15 to 0.69]
  Vaginal Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 7
  Vaginal Biopsy Lysate-Female-Visit 9 |  |  | 0.03 [0.02 to 0.03]
  Vaginal Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Vaginal Biopsy Lysate-Female-Visit 12 |  |  | 0.01 [0.01 to 0.03]
  Vaginal Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 10 | 9 | 7
  Vaginal Biopsy Lysate-Female-Visit 14 | 0.13 [0.07 to 0.38] | 0.87 [0.73 to 1.1] | 0.01 [0.01 to 0.02]
  Vaginal Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 8 | 9 | 0
  Vaginal Biopsy Lysate-Female-Visit 15 | 0.05 [0.02 to 0.06] | 0.11 [0.04 to 0.17] |
  Vaginal Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 7 | 6 | 0
  Vaginal Biopsy Lysate-Female-Visit 16 | 0.01 [0 to 0.01] | 0.03 [0.01 to 0.04] |
  Vaginal Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 5 | 6 | 0
  Vaginal Biopsy Lysate-Female-Visit 17 | 0 [0 to 0] | 0.01 [0 to 0.01] |
  Vaginal Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: IgG-normalized Levels of VRC01 in Genital and Rectal Secretions, as Well as Cervical, Vaginal, and Rectal Tissues (for Groups 1, 2, and 4)
Description: as for outcome 11
Time Frame: Measured through 6 months after the last infusion
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng IgG
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 4: Vaccine
Number analyzed (Participants) | 23 | 23 | 16
pg mAb/ng IgG
  Cervical Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Cervical Biopsy Lysate-Female-Visit 2 | 0.06 [0.02 to 0.09] | 0.02 [0.01 to 0.03] |
  Cervical Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Cervical Biopsy Lysate-Female-Visit 4 |  |  | 25.6 [24.7 to 29.54]
  Cervical Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 5
  Cervical Biopsy Lysate-Female-Visit 5 |  |  | 7.53 [4.5 to 9.92]
  Cervical Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 8
  Cervical Biopsy Lysate-Female-Visit 9 |  |  | 0.99 [0.68 to 1.47]
  Cervical Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Cervical Biopsy Lysate-Female-Visit 12 |  |  | 0.52 [0.19 to 1.12]
  Cervical Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 9 | 9 | 7
  Cervical Biopsy Lysate-Female-Visit 14 | 7.02 [4.52 to 8.53] | 14.6 [10.88 to 20.54] | 0.23 [0.16 to 0.83]
  Cervical Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 9 | 9 | 0
  Cervical Biopsy Lysate-Female-Visit 15 | 0.95 [0.8 to 1.94] | 3.12 [1.39 to 5.05] |
  Cervical Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 7 | 7 | 0
  Cervical Biopsy Lysate-Female-Visit 16 | 0.17 [0.12 to 0.3] | 0.47 [0.34 to 1.32] |
  Cervical Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 6 | 7 | 0
  Cervical Biopsy Lysate-Female-Visit 17 | 0.06 [0.04 to 0.08] | 0.06 [0.04 to 0.08] |
  Cervical Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 7 | 5 | 0
  Rectal Biopsy Lysate-Female-Visit 2 | 0.01 [0.01 to 0.02] | 0.04 [0.01 to 0.4] |
  Rectal Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 9 | 10 | 0
  Rectal Biopsy Lysate-Male-Visit 2 | 0.02 [0.01 to 0.05] | 0.02 [0.01 to 0.04] |
  Rectal Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Rectal Biopsy Lysate-Male-Visit 4 |  |  | 26.33 [22.03 to 32.85]
  Rectal Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 6
  Rectal Biopsy Lysate-Male-Visit 5 |  |  | 6.38 [4.16 to 7.5]
  Rectal Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 7
  Rectal Biopsy Lysate-Male-Visit 9 |  |  | 0.48 [0.35 to 0.94]
  Rectal Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Rectal Biopsy Lysate-Male-Visit 12 |  |  | 0.15 [0.12 to 0.42]
  Rectal Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 6 | 2 | 0
  Rectal Biopsy Lysate-Female-Visit 14 | 9.59 [4.52 to 11.29] | 9.81 [9.46 to 10.16] |
  Rectal Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 5 | 8 | 7
  Rectal Biopsy Lysate-Male-Visit 14 | 10.97 [5.15 to 11.45] | 17.89 [11.6 to 21.82] | 0.07 [0.04 to 0.13]
  Rectal Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 6 | 5 | 0
  Rectal Biopsy Lysate-Female-Visit 15 | 2.1 [1.03 to 2.44] | 1.92 [1.54 to 3.53] |
  Rectal Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 6 | 8 | 0
  Rectal Biopsy Lysate-Male-Visit 15 | 1.07 [0.64 to 1.89] | 4.34 [2.09 to 4.89] |
  Rectal Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 4 | 4 | 0
  Rectal Biopsy Lysate-Female-Visit 16 | 0.32 [0.23 to 0.4] | 0.4 [0.37 to 0.76] |
  Rectal Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 6 | 9 | 0
  Rectal Biopsy Lysate-Male-Visit 16 | 0.07 [0.04 to 0.28] | 0.44 [0.33 to 0.69] |
  Rectal Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 1 | 4 | 0
  Rectal Biopsy Lysate-Female-Visit 17 | 0.1 [0.1 to 0.1] | 0.02 [0.01 to 0.05] |
  Rectal Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 4 | 9 | 0
  Rectal Biopsy Lysate-Male-Visit 17 | 0.02 [0.01 to 0.09] | 0.01 [0.01 to 0.03] |
  Rectal Secretions-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 7
  Rectal Secretions-Male-Visit 1 |  |  | 0.15 [0.12 to 0.29]
  Rectal Secretions-Female-Visit 2: number analyzed (Participants) | 7 | 6 | 0
  Rectal Secretions-Female-Visit 2 | 0.15 [0.11 to 0.34] | 0.23 [0.1 to 0.49] |
  Rectal Secretions-Male-Visit 2: number analyzed (Participants) | 7 | 10 | 0
  Rectal Secretions-Male-Visit 2 | 0.2 [0.09 to 0.3] | 0.09 [0.02 to 0.24] |
  Rectal Secretions-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Female-Visit 4: number analyzed (Participants) | 7 | 6 | 0
  Rectal Secretions-Female-Visit 4 | 2.54 [1.8 to 2.71] | 7.02 [5.19 to 12.83] |
  Rectal Secretions-Male-Visit 4: number analyzed (Participants) | 7 | 8 | 6
  Rectal Secretions-Male-Visit 4 | 2.6 [2.01 to 3.11] | 4.51 [3.66 to 7.49] | 13.07 [8.04 to 15.44]
  Rectal Secretions-Female-Visit 5: number analyzed (Participants) | 6 | 5 | 0
  Rectal Secretions-Female-Visit 5 | 0.39 [0.18 to 0.6] | 1.97 [1.47 to 2.3] |
  Rectal Secretions-Male-Visit 5: number analyzed (Participants) | 7 | 10 | 6
  Rectal Secretions-Male-Visit 5 | 0.78 [0.26 to 0.85] | 1.56 [1.38 to 2.4] | 2.81 [1.68 to 4.13]
  Rectal Secretions-Female-Visit 7: number analyzed (Participants) | 6 | 5 | 0
  Rectal Secretions-Female-Visit 7 | 1.15 [0.48 to 3.03] | 7.63 [6.77 to 8.45] |
  Rectal Secretions-Male-Visit 7: number analyzed (Participants) | 7 | 6 | 6
  Rectal Secretions-Male-Visit 7 | 2.81 [1.61 to 4.5] | 6.46 [6.1 to 7.81] | 1.23 [0.93 to 1.97]
  Rectal Secretions-Female-Visit 9: number analyzed (Participants) | 5 | 5 | 0
  Rectal Secretions-Female-Visit 9 | 0.28 [0.26 to 1.15] | 2.55 [1.49 to 4.69] |
  Rectal Secretions-Male-Visit 9: number analyzed (Participants) | 4 | 7 | 7
  Rectal Secretions-Male-Visit 9 | 0.9 [0.57 to 1.21] | 2.62 [0.97 to 3.17] | 0.18 [0.11 to 0.59]
  Rectal Secretions-Female-Visit 12: number analyzed (Participants) | 3 | 4 | 0
  Rectal Secretions-Female-Visit 12 | 0.89 [0.48 to 0.94] | 2.38 [1.25 to 3.49] |
  Rectal Secretions-Male-Visit 12: number analyzed (Participants) | 4 | 7 | 6
  Rectal Secretions-Male-Visit 12 | 0.9 [0.53 to 1.3] | 1.91 [1.15 to 4.93] | 0.2 [0.15 to 0.38]
  Rectal Secretions-Female-Visit 14: number analyzed (Participants) | 7 | 3 | 0
  Rectal Secretions-Female-Visit 14 | 1.14 [0.47 to 3.82] | 4.81 [2.81 to 9.31] |
  Rectal Secretions-Male-Visit 14: number analyzed (Participants) | 5 | 8 | 6
  Rectal Secretions-Male-Visit 14 | 3.85 [1.55 to 5.4] | 7.18 [3.57 to 9.49] | 0.26 [0.07 to 0.61]
  Rectal Secretions-Female-Visit 15: number analyzed (Participants) | 5 | 5 | 0
  Rectal Secretions-Female-Visit 15 | 0.32 [0.24 to 1.02] | 1.02 [0.97 to 1.26] |
  Rectal Secretions-Male-Visit 15: number analyzed (Participants) | 4 | 5 | 0
  Rectal Secretions-Male-Visit 15 | 0.62 [0.56 to 2.05] | 1.43 [0.57 to 1.95] |
  Rectal Secretions-Female-Visit 16: number analyzed (Participants) | 2 | 4 | 0
  Rectal Secretions-Female-Visit 16 | 0.29 [0.28 to 0.31] | 0.77 [0.39 to 1.19] |
  Rectal Secretions-Male-Visit 16: number analyzed (Participants) | 4 | 7 | 0
  Rectal Secretions-Male-Visit 16 | 0.33 [0.11 to 0.57] | 0.44 [0.33 to 0.71] |
  Rectal Secretions-Female-Visit 17: number analyzed (Participants) | 1 | 3 | 0
  Rectal Secretions-Female-Visit 17 | 2.12 [2.12 to 2.12] | 0.1 [0.07 to 0.56] |
  Rectal Secretions-Male-Visit 17: number analyzed (Participants) | 4 | 7 | 0
  Rectal Secretions-Male-Visit 17 | 0.07 [0.06 to 0.17] | 0.1 [0.05 to 0.13] |
  Semen-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 8
  Semen-Male-Visit 1 |  |  | 0.01 [0.01 to 0.03]
  Semen-Female-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 2: number analyzed (Participants) | 10 | 9 | 0
  Semen-Male-Visit 2 | 0 [0 to 0.01] | 0 [0 to 0.12] |
  Semen-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Semen-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 4: number analyzed (Participants) | 8 | 10 | 8
  Semen-Male-Visit 4 | 5.27 [3.18 to 6.43] | 13.2 [8.94 to 21.71] | 20.07 [15.15 to 23.9]
  Semen-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 5: number analyzed (Participants) | 10 | 10 | 6
  Semen-Male-Visit 5 | 1.88 [0.75 to 2.81] | 5.18 [3.08 to 5.89] | 7.07 [4.96 to 8.52]
  Semen-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 7: number analyzed (Participants) | 9 | 9 | 7
  Semen-Male-Visit 7 | 5.08 [4.52 to 6.58] | 12.66 [9.34 to 22.56] | 2.47 [1.85 to 3.43]
  Semen-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 9: number analyzed (Participants) | 8 | 9 | 7
  Semen-Male-Visit 9 | 1.03 [0.65 to 1.47] | 5.17 [3.35 to 7.28] | 1 [0.65 to 1.52]
  Semen-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 12: number analyzed (Participants) | 7 | 10 | 7
  Semen-Male-Visit 12 | 2.88 [1.53 to 4.37] | 9.72 [6.88 to 10.67] | 0.14 [0.09 to 0.35]
  Semen-Female-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 14: number analyzed (Participants) | 7 | 9 | 7
  Semen-Male-Visit 14 | 5.54 [3.54 to 6.14] | 14.45 [10.11 to 18.05] | 0.06 [0.04 to 0.07]
  Semen-Female-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 15: number analyzed (Participants) | 6 | 9 | 0
  Semen-Male-Visit 15 | 1.47 [0.71 to 2.09] | 3.87 [2.54 to 5.91] |
  Semen-Female-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 16: number analyzed (Participants) | 6 | 10 | 0
  Semen-Male-Visit 16 | 0.17 [0.06 to 0.62] | 0.39 [0.16 to 0.89] |
  Semen-Female-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 17: number analyzed (Participants) | 6 | 9 | 0
  Semen-Male-Visit 17 | 0.01 [0 to 0.01] | 0.01 [0.01 to 0.02] |
  Softcup Fluid-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 5
  Softcup Fluid-Female-Visit 1 |  |  | 0.49 [0.35 to 0.52]
  Softcup Fluid-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 2: number analyzed (Participants) | 6 | 7 | 0
  Softcup Fluid-Female-Visit 2 | 0.04 [0.02 to 0.07] | 0.05 [0.03 to 0.05] |
  Softcup Fluid-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 4: number analyzed (Participants) | 4 | 2 | 5
  Softcup Fluid-Female-Visit 4 | 6.57 [5.87 to 6.6] | 15.26 [13.93 to 16.59] | 14.7 [12.92 to 30.29]
  Softcup Fluid-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 5: number analyzed (Participants) | 4 | 4 | 2
  Softcup Fluid-Female-Visit 5 | 1.35 [0.98 to 2.62] | 5.06 [4.13 to 5.97] | 6.22 [4.18 to 8.26]
  Softcup Fluid-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 7: number analyzed (Participants) | 7 | 6 | 5
  Softcup Fluid-Female-Visit 7 | 4.31 [3.05 to 4.61] | 16.27 [13.22 to 19.9] | 3.75 [1.48 to 3.97]
  Softcup Fluid-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 9: number analyzed (Participants) | 7 | 6 | 4
  Softcup Fluid-Female-Visit 9 | 0.85 [0.66 to 1.34] | 4.78 [4.67 to 5.37] | 1.28 [1.02 to 1.51]
  Softcup Fluid-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 12: number analyzed (Participants) | 2 | 4 | 5
  Softcup Fluid-Female-Visit 12 | 2.45 [2.24 to 2.66] | 9.43 [6.84 to 12.65] | 0.33 [0.17 to 0.44]
  Softcup Fluid-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 14: number analyzed (Participants) | 6 | 6 | 3
  Softcup Fluid-Female-Visit 14 | 6.11 [4.29 to 6.87] | 11.51 [7.2 to 15.3] | 0.14 [0.08 to 0.19]
  Softcup Fluid-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 15: number analyzed (Participants) | 7 | 6 | 0
  Softcup Fluid-Female-Visit 15 | 0.57 [0.51 to 1.03] | 2.05 [0.67 to 3.14] |
  Softcup Fluid-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 16: number analyzed (Participants) | 4 | 4 | 0
  Softcup Fluid-Female-Visit 16 | 0.11 [0.08 to 0.13] | 1.08 [0.53 to 1.54] |
  Softcup Fluid-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 17: number analyzed (Participants) | 4 | 5 | 0
  Softcup Fluid-Female-Visit 17 | 0.09 [0.02 to 0.15] | 0.05 [0.03 to 0.12] |
  Softcup Fluid-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Vaginal Biopsy Lysate-Female-Visit 2 | 0.04 [0.02 to 0.06] | 0.03 [0.02 to 0.04] |
  Vaginal Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Vaginal Biopsy Lysate-Female-Visit 4 |  |  | 25 [20.39 to 34.94]
  Vaginal Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 5
  Vaginal Biopsy Lysate-Female-Visit 5 |  |  | 6.55 [4.74 to 7.79]
  Vaginal Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 7
  Vaginal Biopsy Lysate-Female-Visit 9 |  |  | 0.71 [0.64 to 1.42]
  Vaginal Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Vaginal Biopsy Lysate-Female-Visit 12 |  |  | 0.66 [0.47 to 0.77]
  Vaginal Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 10 | 9 | 7
  Vaginal Biopsy Lysate-Female-Visit 14 | 7.29 [5.29 to 8.13] | 17.29 [11.7 to 24.46] | 0.2 [0.17 to 0.58]
  Vaginal Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 8 | 9 | 0
  Vaginal Biopsy Lysate-Female-Visit 15 | 1 [0.85 to 1.43] | 2.67 [1.51 to 4.85] |
  Vaginal Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 7 | 6 | 0
  Vaginal Biopsy Lysate-Female-Visit 16 | 0.21 [0.16 to 0.32] | 0.56 [0.29 to 1.71] |
  Vaginal Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 5 | 6 | 0
  Vaginal Biopsy Lysate-Female-Visit 17 | 0.03 [0.01 to 0.04] | 0.06 [0.03 to 0.08] |
  Vaginal Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0

15. Primary Outcome: Protein-normalized Levels of VRC01 in Genital and Rectal Secretions, as Well as Cervical, Vaginal, and Rectal Tissues (for Groups 1, 2, and 4)
Description: as for outcome 12
Time Frame: Measured through 6 months after the last infusion
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng total protein
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 4: Vaccine
Number analyzed (Participants) | 23 | 23 | 16
pg mAb/ng total protein
  Cervical Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Cervical Biopsy Lysate-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Cervical Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Cervical Biopsy Lysate-Female-Visit 4 |  |  | 1.12 [0.93 to 1.26]
  Cervical Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 5
  Cervical Biopsy Lysate-Female-Visit 5 |  |  | 0.24 [0.23 to 0.26]
  Cervical Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 8
  Cervical Biopsy Lysate-Female-Visit 9 |  |  | 0.04 [0.03 to 0.05]
  Cervical Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Cervical Biopsy Lysate-Female-Visit 12 |  |  | 0.02 [0.01 to 0.03]
  Cervical Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 9 | 9 | 7
  Cervical Biopsy Lysate-Female-Visit 14 | 0.3 [0.26 to 0.48] | 0.87 [0.84 to 0.96] | 0.01 [0.01 to 0.03]
  Cervical Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 9 | 9 | 0
  Cervical Biopsy Lysate-Female-Visit 15 | 0.05 [0.04 to 0.1] | 0.16 [0.1 to 0.22] |
  Cervical Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 7 | 7 | 0
  Cervical Biopsy Lysate-Female-Visit 16 | 0.01 [0.01 to 0.02] | 0.03 [0.01 to 0.05] |
  Cervical Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Cervical Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 6 | 7 | 0
  Cervical Biopsy Lysate-Female-Visit 17 | 0 [0 to 0.01] | 0 [0 to 0] |
  Cervical Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 7 | 5 | 0
  Rectal Biopsy Lysate-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0.01] |
  Rectal Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 9 | 10 | 0
  Rectal Biopsy Lysate-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Rectal Biopsy Lysate-Male-Visit 4 |  |  | 0.41 [0.3 to 0.53]
  Rectal Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 6
  Rectal Biopsy Lysate-Male-Visit 5 |  |  | 0.08 [0.06 to 0.12]
  Rectal Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 7
  Rectal Biopsy Lysate-Male-Visit 9 |  |  | 0.01 [0.01 to 0.02]
  Rectal Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Rectal Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Rectal Biopsy Lysate-Male-Visit 12 |  |  | 0 [0 to 0.01]
  Rectal Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 6 | 2 | 0
  Rectal Biopsy Lysate-Female-Visit 14 | 0.13 [0.09 to 0.18] | 0.17 [0.16 to 0.19] |
  Rectal Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 5 | 8 | 7
  Rectal Biopsy Lysate-Male-Visit 14 | 0.1 [0.07 to 0.17] | 0.23 [0.2 to 0.39] | 0 [0 to 0]
  Rectal Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 6 | 5 | 0
  Rectal Biopsy Lysate-Female-Visit 15 | 0.03 [0.02 to 0.04] | 0.04 [0.03 to 0.04] |
  Rectal Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 6 | 8 | 0
  Rectal Biopsy Lysate-Male-Visit 15 | 0.02 [0.01 to 0.03] | 0.06 [0.05 to 0.1] |
  Rectal Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 4 | 4 | 0
  Rectal Biopsy Lysate-Female-Visit 16 | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.02] |
  Rectal Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 6 | 9 | 0
  Rectal Biopsy Lysate-Male-Visit 16 | 0 [0 to 0.01] | 0.01 [0 to 0.02] |
  Rectal Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 1 | 4 | 0
  Rectal Biopsy Lysate-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 4 | 9 | 0
  Rectal Biopsy Lysate-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 7
  Rectal Secretions-Male-Visit 1 |  |  | 0 [0 to 0]
  Rectal Secretions-Female-Visit 2: number analyzed (Participants) | 7 | 6 | 0
  Rectal Secretions-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 2: number analyzed (Participants) | 7 | 10 | 0
  Rectal Secretions-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Rectal Secretions-Female-Visit 4: number analyzed (Participants) | 7 | 6 | 0
  Rectal Secretions-Female-Visit 4 | 0.01 [0 to 0.01] | 0 [0 to 0.01] |
  Rectal Secretions-Male-Visit 4: number analyzed (Participants) | 7 | 8 | 6
  Rectal Secretions-Male-Visit 4 | 0.01 [0 to 0.01] | 0.03 [0 to 0.06] | 0.02 [0.01 to 0.04]
  Rectal Secretions-Female-Visit 5: number analyzed (Participants) | 6 | 5 | 0
  Rectal Secretions-Female-Visit 5 | 0 [0 to 0] | 0.01 [0 to 0.04] |
  Rectal Secretions-Male-Visit 5: number analyzed (Participants) | 7 | 10 | 6
  Rectal Secretions-Male-Visit 5 | 0 [0 to 0] | 0.01 [0.01 to 0.01] | 0 [0 to 0.01]
  Rectal Secretions-Female-Visit 7: number analyzed (Participants) | 6 | 5 | 0
  Rectal Secretions-Female-Visit 7 | 0 [0 to 0] | 0.01 [0.01 to 0.02] |
  Rectal Secretions-Male-Visit 7: number analyzed (Participants) | 7 | 6 | 6
  Rectal Secretions-Male-Visit 7 | 0.01 [0 to 0.01] | 0.03 [0.02 to 0.1] | 0 [0 to 0.01]
  Rectal Secretions-Female-Visit 9: number analyzed (Participants) | 5 | 5 | 0
  Rectal Secretions-Female-Visit 9 | 0 [0 to 0] | 0.01 [0 to 0.01] |
  Rectal Secretions-Male-Visit 9: number analyzed (Participants) | 4 | 7 | 7
  Rectal Secretions-Male-Visit 9 | 0 [0 to 0.01] | 0 [0 to 0.06] | 0 [0 to 0]
  Rectal Secretions-Female-Visit 12: number analyzed (Participants) | 3 | 4 | 0
  Rectal Secretions-Female-Visit 12 | 0 [0 to 0] | 0 [0 to 0.01] |
  Rectal Secretions-Male-Visit 12: number analyzed (Participants) | 4 | 7 | 6
  Rectal Secretions-Male-Visit 12 | 0 [0 to 0.01] | 0.01 [0 to 0.02] | 0 [0 to 0]
  Rectal Secretions-Female-Visit 14: number analyzed (Participants) | 7 | 3 | 0
  Rectal Secretions-Female-Visit 14 | 0 [0 to 0.02] | 0.01 [0.01 to 0.01] |
  Rectal Secretions-Male-Visit 14: number analyzed (Participants) | 5 | 8 | 6
  Rectal Secretions-Male-Visit 14 | 0.01 [0 to 0.08] | 0.01 [0 to 0.03] | 0 [0 to 0]
  Rectal Secretions-Female-Visit 15: number analyzed (Participants) | 5 | 5 | 0
  Rectal Secretions-Female-Visit 15 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 15: number analyzed (Participants) | 4 | 5 | 0
  Rectal Secretions-Male-Visit 15 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Female-Visit 16: number analyzed (Participants) | 2 | 4 | 0
  Rectal Secretions-Female-Visit 16 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 16: number analyzed (Participants) | 4 | 7 | 0
  Rectal Secretions-Male-Visit 16 | 0 [0 to 0] | 0 [0 to 0.01] |
  Rectal Secretions-Female-Visit 17: number analyzed (Participants) | 1 | 3 | 0
  Rectal Secretions-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Rectal Secretions-Male-Visit 17: number analyzed (Participants) | 4 | 7 | 0
  Rectal Secretions-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Semen-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 8
  Semen-Male-Visit 1 |  |  | 0 [0 to 0]
  Semen-Female-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 2: number analyzed (Participants) | 10 | 9 | 0
  Semen-Male-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Semen-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Semen-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 4: number analyzed (Participants) | 8 | 10 | 8
  Semen-Male-Visit 4 | 0.01 [0 to 0.01] | 0.02 [0.02 to 0.05] | 0.02 [0.02 to 0.02]
  Semen-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 5: number analyzed (Participants) | 10 | 10 | 6
  Semen-Male-Visit 5 | 0 [0 to 0] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01]
  Semen-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 7: number analyzed (Participants) | 9 | 9 | 7
  Semen-Male-Visit 7 | 0.01 [0 to 0.01] | 0.02 [0.02 to 0.03] | 0 [0 to 0]
  Semen-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 9: number analyzed (Participants) | 8 | 9 | 7
  Semen-Male-Visit 9 | 0 [0 to 0] | 0.01 [0.01 to 0.02] | 0 [0 to 0]
  Semen-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 12: number analyzed (Participants) | 7 | 10 | 7
  Semen-Male-Visit 12 | 0 [0 to 0] | 0.02 [0.01 to 0.03] | 0 [0 to 0]
  Semen-Female-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 14: number analyzed (Participants) | 7 | 9 | 7
  Semen-Male-Visit 14 | 0 [0 to 0.01] | 0.02 [0.02 to 0.03] | 0 [0 to 0]
  Semen-Female-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 15: number analyzed (Participants) | 6 | 9 | 0
  Semen-Male-Visit 15 | 0 [0 to 0] | 0.01 [0 to 0.02] |
  Semen-Female-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 16: number analyzed (Participants) | 6 | 10 | 0
  Semen-Male-Visit 16 | 0 [0 to 0] | 0 [0 to 0] |
  Semen-Female-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Semen-Male-Visit 17: number analyzed (Participants) | 6 | 9 | 0
  Semen-Male-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Softcup Fluid-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 5
  Softcup Fluid-Female-Visit 1 |  |  | 0.01 [0.01 to 0.02]
  Softcup Fluid-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 2: number analyzed (Participants) | 6 | 7 | 0
  Softcup Fluid-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Softcup Fluid-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 4: number analyzed (Participants) | 4 | 2 | 5
  Softcup Fluid-Female-Visit 4 | 0.29 [0.18 to 0.44] | 0.68 [0.54 to 0.82] | 0.96 [0.5 to 1.03]
  Softcup Fluid-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 5: number analyzed (Participants) | 4 | 4 | 2
  Softcup Fluid-Female-Visit 5 | 0.03 [0.02 to 0.06] | 0.16 [0.14 to 0.22] | 0.19 [0.18 to 0.21]
  Softcup Fluid-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 7: number analyzed (Participants) | 7 | 6 | 5
  Softcup Fluid-Female-Visit 7 | 0.21 [0.19 to 0.26] | 0.8 [0.57 to 0.95] | 0.07 [0.04 to 0.09]
  Softcup Fluid-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 9: number analyzed (Participants) | 7 | 6 | 4
  Softcup Fluid-Female-Visit 9 | 0.04 [0.04 to 0.06] | 0.23 [0.22 to 0.26] | 0.04 [0.04 to 0.06]
  Softcup Fluid-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 12: number analyzed (Participants) | 2 | 4 | 5
  Softcup Fluid-Female-Visit 12 | 0.28 [0.24 to 0.32] | 0.54 [0.41 to 0.57] | 0.01 [0.01 to 0.01]
  Softcup Fluid-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 14: number analyzed (Participants) | 6 | 6 | 3
  Softcup Fluid-Female-Visit 14 | 0.29 [0.25 to 0.33] | 0.49 [0.43 to 0.73] | 0 [0 to 0.01]
  Softcup Fluid-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 15: number analyzed (Participants) | 7 | 6 | 0
  Softcup Fluid-Female-Visit 15 | 0.06 [0.03 to 0.08] | 0.07 [0.02 to 0.13] |
  Softcup Fluid-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 16: number analyzed (Participants) | 4 | 4 | 0
  Softcup Fluid-Female-Visit 16 | 0.01 [0.01 to 0.01] | 0.03 [0.01 to 0.07] |
  Softcup Fluid-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Softcup Fluid-Female-Visit 17: number analyzed (Participants) | 4 | 5 | 0
  Softcup Fluid-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0] |
  Softcup Fluid-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 1: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 2: number analyzed (Participants) | 13 | 13 | 0
  Vaginal Biopsy Lysate-Female-Visit 2 | 0 [0 to 0] | 0 [0 to 0] |
  Vaginal Biopsy Lysate-Male-Visit 2: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 3: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 4: number analyzed (Participants) | 0 | 0 | 8
  Vaginal Biopsy Lysate-Female-Visit 4 |  |  | 0.86 [0.59 to 1.1]
  Vaginal Biopsy Lysate-Male-Visit 4: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 5: number analyzed (Participants) | 0 | 0 | 5
  Vaginal Biopsy Lysate-Female-Visit 5 |  |  | 0.25 [0.14 to 0.31]
  Vaginal Biopsy Lysate-Male-Visit 5: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Male-Visit 7: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 9: number analyzed (Participants) | 0 | 0 | 7
  Vaginal Biopsy Lysate-Female-Visit 9 |  |  | 0.03 [0.02 to 0.04]
  Vaginal Biopsy Lysate-Male-Visit 9: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 12: number analyzed (Participants) | 0 | 0 | 7
  Vaginal Biopsy Lysate-Female-Visit 12 |  |  | 0.01 [0.01 to 0.02]
  Vaginal Biopsy Lysate-Male-Visit 12: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 14: number analyzed (Participants) | 10 | 9 | 7
  Vaginal Biopsy Lysate-Female-Visit 14 | 0.21 [0.14 to 0.32] | 0.76 [0.7 to 0.82] | 0.01 [0 to 0.02]
  Vaginal Biopsy Lysate-Male-Visit 14: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 15: number analyzed (Participants) | 8 | 9 | 0
  Vaginal Biopsy Lysate-Female-Visit 15 | 0.04 [0.03 to 0.05] | 0.11 [0.07 to 0.14] |
  Vaginal Biopsy Lysate-Male-Visit 15: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 16: number analyzed (Participants) | 7 | 6 | 0
  Vaginal Biopsy Lysate-Female-Visit 16 | 0.01 [0.01 to 0.01] | 0.02 [0.01 to 0.05] |
  Vaginal Biopsy Lysate-Male-Visit 16: number analyzed (Participants) | 0 | 0 | 0
  Vaginal Biopsy Lysate-Female-Visit 17: number analyzed (Participants) | 5 | 6 | 0
  Vaginal Biopsy Lysate-Female-Visit 17 | 0 [0 to 0] | 0 [0 to 0.01] |
  Vaginal Biopsy Lysate-Male-Visit 17: number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Ex Vivo Inhibition of HIV-1 Infectivity in Tissue Biopsies (for Groups 1, 2, and 3)
Description: Magnitudes of ex vivo HIV-1 infection were measured by the tissue luminescence assay (TLA). Susceptibility to viral infection in the ex vivo challenge assay is summarized by the area under the viral infectivity curve (AUC) based on log-transformed RLU values between 3-21 days of culture, indicated as AUCday3-21.
Time Frame: Cervical biopsies collected at visits 2 and 14; Rectal biopsies collected at visits 2, 14, 15, 16, 17, 18, 19 (19 not apply for Du422.1); Vaginal biopsies collected at visits 2 and 14, 15, 16, 17. RLU measured every 3 days, during culture days 3-21.
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Log(RLU)*Day
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine
Number analyzed (Participants) | 23 | 23 | 7
Log(RLU)*Day
  Cervical Biopsy-Bal26-visit 2: number analyzed (Participants) | 11 | 12 | 3
  Cervical Biopsy-Bal26-visit 2 | 134.61 [114.47 to 138.29] | 128.69 [120.23 to 132.74] | 125.66 [120.08 to 136.16]
  Cervical Biopsy-Bal26-visit 14: number analyzed (Participants) | 10 | 10 | 2
  Cervical Biopsy-Bal26-visit 14 | 81.74 [80.14 to 89.01] | 80.03 [78.51 to 80.27] | 82.33 [81.61 to 83.05]
  Rectal Biopsy-1086-visit 2: number analyzed (Participants) | 16 | 15 | 5
  Rectal Biopsy-1086-visit 2 | 149.47 [145.48 to 152.04] | 151.28 [144.06 to 153.78] | 145.97 [134.13 to 150.66]
  Rectal Biopsy-1086-visit 14: number analyzed (Participants) | 10 | 14 | 5
  Rectal Biopsy-1086-visit 14 | 147.95 [145.12 to 150.71] | 147.69 [141.98 to 151.35] | 152.22 [150.83 to 152.75]
  Rectal Biopsy-1086-visit 15: number analyzed (Participants) | 11 | 14 | 5
  Rectal Biopsy-1086-visit 15 | 150.66 [143.88 to 158.18] | 148.86 [137.49 to 152.6] | 145.42 [139.31 to 147.3]
  Rectal Biopsy-1086-visit 16: number analyzed (Participants) | 10 | 14 | 5
  Rectal Biopsy-1086-visit 16 | 147.24 [144.16 to 151.24] | 145.82 [142.66 to 151.74] | 153.31 [146.73 to 153.45]
  Rectal Biopsy-1086-visit 17: number analyzed (Participants) | 8 | 12 | 4
  Rectal Biopsy-1086-visit 17 | 147.56 [138.79 to 150.2] | 148.37 [146.89 to 150.47] | 148.82 [136.03 to 154.05]
  Rectal Biopsy-1086-visit 18: number analyzed (Participants) | 0 | 0 | 2
  Rectal Biopsy-1086-visit 18 |  |  | 139.29 [133.19 to 145.38]
  Rectal Biopsy-1086-visit 19: number analyzed (Participants) | 0 | 0 | 1
  Rectal Biopsy-1086-visit 19 |  |  | 148.87 [148.87 to 148.87]
  Rectal Biopsy-Bal26-visit 2: number analyzed (Participants) | 16 | 15 | 5
  Rectal Biopsy-Bal26-visit 2 | 142.83 [139.27 to 144.63] | 139.99 [136.37 to 144.52] | 140.62 [140.35 to 140.69]
  Rectal Biopsy-Bal26-visit 14: number analyzed (Participants) | 11 | 14 | 5
  Rectal Biopsy-Bal26-visit 14 | 93.17 [90.26 to 96.57] | 97.41 [89.65 to 107.71] | 90.31 [88.38 to 91.73]
  Rectal Biopsy-Bal26-visit 15: number analyzed (Participants) | 11 | 14 | 5
  Rectal Biopsy-Bal26-visit 15 | 136.16 [107.58 to 144.78] | 117.51 [105.53 to 137.13] | 89.36 [88.87 to 97.36]
  Rectal Biopsy-Bal26-visit 16: number analyzed (Participants) | 12 | 14 | 5
  Rectal Biopsy-Bal26-visit 16 | 136.69 [130.48 to 142.45] | 135.71 [127.26 to 144.7] | 92.33 [88.39 to 114.91]
  Rectal Biopsy-Bal26-visit 17: number analyzed (Participants) | 8 | 12 | 4
  Rectal Biopsy-Bal26-visit 17 | 138.8 [135.35 to 143.92] | 140.59 [137.3 to 143.16] | 129.17 [105.55 to 140.14]
  Rectal Biopsy-Bal26-visit 18: number analyzed (Participants) | 0 | 0 | 2
  Rectal Biopsy-Bal26-visit 18 |  |  | 115.21 [91.07 to 139.34]
  Rectal Biopsy-Bal26-visit 19: number analyzed (Participants) | 0 | 0 | 1
  Rectal Biopsy-Bal26-visit 19 |  |  | 106.05 [106.05 to 106.05]
  Rectal Biopsy-Du422.1-visit 2: number analyzed (Participants) | 14 | 12 | 5
  Rectal Biopsy-Du422.1-visit 2 | 141.44 [129.25 to 150.08] | 142.74 [127.52 to 145.48] | 151.14 [146.98 to 152.85]
  Rectal Biopsy-Du422.1-visit 14: number analyzed (Participants) | 7 | 12 | 4
  Rectal Biopsy-Du422.1-visit 14 | 145.48 [137.7 to 155.83] | 138.99 [131.85 to 143.72] | 143.46 [129.24 to 151.88]
  Rectal Biopsy-Du422.1-visit 15: number analyzed (Participants) | 8 | 11 | 4
  Rectal Biopsy-Du422.1-visit 15 | 141.14 [123.53 to 147.23] | 139.5 [123.33 to 148.93] | 145.45 [140.12 to 149.79]
  Rectal Biopsy-Du422.1-visit 16: number analyzed (Participants) | 8 | 11 | 4
  Rectal Biopsy-Du422.1-visit 16 | 143.53 [139.83 to 147.13] | 142 [139.9 to 148.63] | 144.16 [138.03 to 149.44]
  Rectal Biopsy-Du422.1-visit 17: number analyzed (Participants) | 5 | 4 | 3
  Rectal Biopsy-Du422.1-visit 17 | 145.72 [138.63 to 149.71] | 139.58 [133.97 to 145.52] | 150.64 [147.97 to 152.59]
  Rectal Biopsy-Du422.1-visit 18: number analyzed (Participants) | 0 | 0 | 1
  Rectal Biopsy-Du422.1-visit 18 |  |  | 130.75 [130.75 to 130.75]
  Vaginal Biopsy-Bal26-visit 2: number analyzed (Participants) | 13 | 12 | 3
  Vaginal Biopsy-Bal26-visit 2 | 128.69 [127.25 to 135.46] | 130.33 [122.46 to 140.45] | 116.62 [81.53 to 140.27]
  Vaginal Biopsy-Bal26-visit 14: number analyzed (Participants) | 11 | 10 | 2
  Vaginal Biopsy-Bal26-visit 14 | 80.78 [78.33 to 88.97] | 82.89 [80.98 to 92.99] | 80.88 [79.45 to 82.32]
  Vaginal Biopsy-Bal26-visit 15: number analyzed (Participants) | 10 | 9 | 3
  Vaginal Biopsy-Bal26-visit 15 | 94.41 [81.3 to 109.8] | 89.85 [81.33 to 105.55] | 82.26 [80.61 to 83.04]
  Vaginal Biopsy-Bal26-visit 16: number analyzed (Participants) | 9 | 8 | 3
  Vaginal Biopsy-Bal26-visit 16 | 128.28 [118.47 to 132.88] | 104.97 [93.97 to 112.99] | 82.76 [79.37 to 83.01]
  Vaginal Biopsy-Bal26-visit 17: number analyzed (Participants) | 1 | 2 | 0
  Vaginal Biopsy-Bal26-visit 17 | 131.37 [131.37 to 131.37] | 137.49 [130.71 to 144.27] |

ADVERSE EVENTS:
Time Frame: Measured through participant's last study visit, at 6 months to 1 1/2 years after study entry (depending on which group participants are in)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Pre-treatment
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/7 | 0/16 | 0/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/23 | 1/7 | 0/16 | 1/10 | 0/1
Other Adverse Events (participants affected / at risk) | 22/23 | 18/23 | 7/7 | 7/16 | 3/10 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=23) | Group 2: Vaccine (N=23) | Group 3: Vaccine (N=7) | Group 4: Vaccine (N=16) | Group 5: Vaccine (N=10) | Group 6: Pre-treatment (N=1)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=23) | Group 2: Vaccine (N=23) | Group 3: Vaccine (N=7) | Group 4: Vaccine (N=16) | Group 5: Vaccine (N=10) | Group 6: Pre-treatment (N=1)
Any Event in SOC (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 7 (10) | 6 (13) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Infections and infestations) | 16 (37) | 17 (31) | 7 (12) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida cervicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoid infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (13) | 9 (15) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 7 (8) | 3 (6) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 9 (22) | 10 (16) | 3 (8) | 2 (5) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 6 (11) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystadenofibroma of fallopian tube (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 5 (5) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 6 (13) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulva cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 6 (9) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02797171/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT02797171/SAP_001.pdf